CLINICAL TRIAL: NCT06000033
Title: Combination of Disitamab Vedotin and Anlotinib in the Treatment of HR-Negative, HER2-Low-Expressing Metastatic Breast Cancer: A Single-Arm, Multicenter, Phase II Clinical Study
Brief Title: Study of Disitamab Vedotin and Anlotinib in Patients With HR-Negative, HER2-Low-Expressing Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48HR-/HER2LOW
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
Keywords: HER2 low expression; Breast Cancer; RC48; Disitamab Vedotin
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48+Anlotinib (Experimental): Disitamab Vedotin : 2 mg/kg，ivgtt，d1-14/28day/cycle Anlotinib: 12mg once daily (taken before meals) orally, continuously for 2 weeks followed by a 1-week break. Each cycle consists of 21 days.
  Interventions: Drug: Disitamab Vedotin+Anlotinib

INTERVENTIONS:
Drug: Disitamab Vedotin+Anlotinib — Disitamab Vedotin:2 mg/kg，ivgtt，d1-14/28day/cycle Anlotinib: 12mg once daily (taken before meals) orally, continuously for 2 weeks followed by a 1-week break. Each cycle consists of 21 days.

SUMMARY:
Disitamab Vedotin (RC48) contains the novel humanized anti-HER2 antibody conjugated to monomethyl auristatin E (MMAE) via a cleavable linker , which is the first ADC drug that was independently developed by Rongchang Biology .The aim of this study is to evaluate the efficacy and safety of RC48 in Combination with Anlotinib for the treatment of metastatic breast cancer with HR negativity and HER2 low expression.

ELIGIBILITY:
Inclusion Criteria:

* 1)At the time of signing the informed consent form, the age is ≥ 18 years old, regardless of gender;
* 2)Patients with pathohistologically proven, locally advanced or metastatic breast cancer have progressed through second-line standard treatment;
* 3)The immunohistochemical (IHC) test results of archived tissue (within 6 months) or fresh biopsy lesions were negative for ER and PR, while patients with low HER-2 expression were HR -, HER2IHC1+, or HER2IHC2+and ISH negative;
* 4)ECOGPS: 0-1 points;
* 5)Expected survival time>12 weeks;
* 6)Adequate organ function: bone marrow function: hemoglobin ≥ 9g/dL; Absolute neutrophil count ≥ 1.5 × 109/L; White blood cell count ≥ 3.0 × 109/L; Platelets ≥ 100 × 109/L; Liver function: serum total bilirubin ≤ 1.5 times the upper limit of normal value (ULN); Aspartic acid Transaminase (AST) and alanine Transaminase (ALT) ≤ 3.0 × ULN (or ≤ 5.0 in the presence of liver metastasis) × ULN) Renal function: blood creatinine ≤ 1.5 × The creatinine clearance rate (CrCl) calculated by ULN or Cockcroft Fault formula method is ≥ 60mL/min; Cardiac function: New York Heart Association (NYHA) grading<3; Left ventricular Ejection fraction ≥ 50%;
* 7)At least one measurable lesion defined in RECIST version 1.1;
* 8)Women of childbearing age must have taken reliable contraceptive measures or conducted a Pregnancy test (serum or urine) within 7 days before enrollment, and the result is negative, and are willing to use appropriate methods of contraception during the test and 8 weeks after the last administration of the test drug. For males, it is necessary to agree to use appropriate methods of contraception or undergo surgical sterilization during the trial period and 8 weeks after the last administration of the investigational drug;
* 9)The subjects voluntarily joined this study and signed an informed consent form, with good compliance and cooperation in follow-up.

Exclusion Criteria:

* 1)The second-line treatment within 3 months is paclitaxel drug therapy;
* 2)Received antitumor therapy or radiation therapy for any malignancy within the previous five years, excluding cured cervical carcinoma in situ, skin basal cell carcinoma, or squamous cell carcinoma;
* 3)had a major non-breast cancer related surgery in the 4 weeks prior to enrollment, or had not fully recovered from such surgery;
* 4)Previously received ADC drugs, anti-angiogenesis drugs, anti-HER2 and other treatments;
* 5)Serious cardiovascular and cerebrovascular disease or discomfort, including but not limited to the following diseases: - History of confirmed heart failure or systolic dysfunction (LVEF<50%) - high-risk uncontrolled arrhythmias - angina, acute myocardial infarction - clinically significant valvular heart disease - poorly controlled hypertension (systolic blood pressure >180mmHg and/or diastolic blood pressure >100mmHg)
* 6)known allergic history of the drug components of this protocol;
* 7)A history of immunodeficiency, including HIV testing positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
* 8)symptomatic brain metastases or brain metastases (excluding prophylactic cranial irradiation) within 4 weeks prior to initiation of treatment; 9) Pregnant and lactating women, fertile women who tested positive for baseline pregnancy tests, or patients of childbearing age who were unwilling to take effective contraception throughout the trial period;
* 9)Have a serious concomitant condition or other comorbid condition that interferes with planned treatment, or any other condition in which the investigator deems the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-08-10 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 1year
  The percentage of cases that have achieved complete or partial remission after drug treatment compared to the total evaluable cases.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 2years
  All adverse events (AEs) in this study will be encoded using MedDRA and classified according to the NCICTCAEv5.0 grading system.
Overall Survival (OS) | 2years
  Defined as the time from the beginning of the patient's treatment to death from any cause.
Disease Control Rate (DCR) | 1year
  The proportion of patients who achieve complete remission (CR), partial remission (PR), or disease stability (SD) during or after treatment
Duration of Response (DOR) | 1year
  Defined as the date from which tumor remission was first recorded (evaluated according to the RECIST 1.1 standard) to the date when disease progression was first recorded (evaluated according to the RECIST 1.1 standard) or the date of death from any cause.
AEs | 2years
  All adverse events (AEs) in this study will be encoded using MedDRA and classified according to the NCICTCAEv5.0 grading system.

IPD SHARING:
Plan to Share IPD: No